CLINICAL TRIAL: NCT02854189
Title: Department of Orthopaedics Faculty of Medicine Thammasat University Thailand
Brief Title: The Results of Oxford Unicompartmental Knee Arthroplasty in Patients With and Without Preoperative Genu Recurvatum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Boonchana Pongcharoen, Principal investigator, Thammasat University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MTU-EC-OT-0-051/59
Record Dates: First submitted 2016-06-06; First posted 2016-08-03 (Estimated); Last update posted 2020-06-04 (Actual); Status verified 2016-07

CONDITIONS: Primary Gonarthrosis; Genu Recurvatum

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- patients with genu recurvatum (Other): The medial osteoarthritis knees with genu recurvatum were included in this study. Patients had been treated with cemented minimally invasive surgery Oxford unicompartmental knee arthroplasty and had had a minimum of 24 months of follow-up.The incidence of postoperative genu recurvatum, postoperative hyperextension angle, and the knee society score were recorded.
  Interventions: Device: Oxford unicompartmental knee arthroplasty
- patients without genu recurvatum (Other): The medial osteoarthritis knees without genu recurvatum were included in this study. Patients had been treated with cemented minimally invasive surgery Oxford unicompartmental knee arthroplasty and had had a minimum of 24 months of follow-up.The incidence of postoperative genu recurvatum, postoperative hyperextension angle, and the knee society score were recorded.
  Interventions: Device: Oxford unicompartmental knee arthroplasty

INTERVENTIONS:
Device: Oxford unicompartmental knee arthroplasty — The Oxford unicompartmental knee arthroplasty was applied in all patients with medial osteoarthritis knee.The Oxford unicompartmental knee arthroplasty is mobile bearing unicompartmental knee arthroplasty.

SUMMARY:
The purpose of this study is to explore the effects of the Oxford unicompartmental knee arthroplasty on two groups of patients, namely one with genu recurvatum before the procedure and one without. Specifically, this study compare the number of occurrences of postoperative genu recurvatum and the postoperative hyperextension angles among the patients. Additionally, the knee scores, the pain scores, and the functional scores for the two groups of patients are compared.

Materials and methods: This study prospectively followed 104 patients (114 knees) who had been treated with cemented minimally invasive surgery unicompartmental knee arthroplasty and had had a minimum of 24 months of follow-up. The patients were divided into two groups: those without preoperative genu recurvatum (85 patients; 94 knees) and those with preoperative genu recurvatum (19 patients; 20 knees). The incidence of the postoperative genu recurvatum, the postoperative hyperextension angles, the knee scores, the pain scores, and the functional scores were recorded and compared between two groups..

DETAILED DESCRIPTION:
The patients in both groups were applied with cemented Oxford unicompartmental knee arthroplasty with the same surgeon. The all patients were performed surgery with minimally invasive surgery technique. The gender, site, range of motion, alignment of prosthesis, operative time, blood loss, and posterior slope of tibial component also were recorded and compared between two groups. The incidence of postoperative genu recurvatum, gender, and site were computed using Fisher's exact test. The hyperextension angle, knee score, pain score, functional score,range of motion, alignment of prosthesis, posterior slope of tibial component, operative time, and blood loss were compared with student t-test.

ELIGIBILITY:
Inclusion Criteria:

* The medial OA knee with older than 40 years of age, ROM greater than 90°, varus deformity less than 25°, and flexion contractures less than 20°

Exclusion Criteria:

* patients who were diagnosed spontaneous osteonecrosis of knee (SPONK), patients with intraoperative ACL insufficiency, post traumatic arthritis, gouty arthritis, inflammatory joints.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2011-01; Primary Completion 2013-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
hyperextension angle, the incidence of postoperative genu recurvatum | 2 years
  hyperextension angle, the incidence of postoperative genu recurvatum

IPD SHARING:
Plan to Share IPD: No